CLINICAL TRIAL: NCT06089109
Title: Violence Intervention and Prevention (VIP) Corps to Reduce Maternal Injuries and Deaths Due to Violence
Brief Title: Creating VIP Corps to Reduce Maternal Deaths
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann Coker (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ann Coker, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 77241; 5 ASTWH210102-02-00 (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2023-09-29; First posted 2023-10-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Maternal Morbidity and Mortality
Keywords: Maternal Morbidity; Maternal Mortality; VIP Corps; Pregnancy-associated injuries; Pregnancy-associated deaths
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maternal Injury and Death Intervention (Experimental): Our research team created a VIP Corps online, interactive learning management system (LMS) training. This VIP Corps online training will be offered to students enrolled in a helping profession. Students are randomized to this experimental intervention arm. This training seeks to provide helping professionals with information and resources to identify, intervene, and prevent maternal injuries from interpersonal violence, substance use/disorder (IPV and SU/D). This training will provide students with the knowledge, skills, and efficacy to intervene and build capacity for prevention of maternal injuries and death due to violence.
  Interventions: Behavioral: Implementation and Effectiveness of VIP Corps Training
- Development of a Maternal Injury Surveillance System (Active Comparator): Proposal of a novel Maternal Injury Surveillance System (MISS) as a complement to the existing maternal mortality surveillance available within Kentucky Violent Death Reporting System (KVDRS)
  Interventions: Behavioral: The Big 3

INTERVENTIONS:
Behavioral: The Big 3 — Our research team has developed an online, interactive learning management system (LMS) training. This training seeks to provide helping professionals with information and resources to identify, intervene, and prevent maternal injuries from interpersonal violence, substance use/disorder (IPV and SU/D). This training will provide healthcare professionals with the knowledge, skills, and efficacy to intervene and build capacity for prevention of maternal injuries and death due to violence.
  Arms: Development of a Maternal Injury Surveillance System
Behavioral: Implementation and Effectiveness of VIP Corps Training — Implement and evaluate the effectiveness of VIP Corps training aimed at students enrolled in helping professions in their last program year. intervention efficacy to change in students' knowledge, attitudes, and practices of intimate partner violence (IPV) screening, detection, and referrals; participant practices will be the primary, longer-term outcome; while changes in knowledge and attitudes will be short-term outcomes. Secondary outcomes will include changes in detecting symptoms of a) SU/D and b) depression and/or anxiety and providing appropriate resources.
  Arms: Maternal Injury and Death Intervention

SUMMARY:
The goal of this observational study is to create and rigorously evaluate a violence intervention and prevention corps (VIP Corps) training using a randomized controlled trial among undergraduate and professional students; and to develop a novel maternal injury surveillance system (MISS) to complement an existing maternal violent death registry in Kentucky.

DETAILED DESCRIPTION:
The participant population defined in this study are undergraduate and professional students within their last educational year in a helping professionals program at the University of Kentucky, ages 18-30. This study will permit the creation of effective programming to train the next generation of health and social service professionals prepared to help reduce Kentucky's maternal mortality and injury rates over time with implementation.

Aim 1:

1. Create and rigorously evaluating Violence Intervention and Prevention Corps (VIP Corps) training using a randomized controlled trial among undergraduate and professional students.
2. Develop a novel maternal injury surveillance system (MISS) as a complement to an existing maternal violent deaths registry to accurately and reliably enumerate maternal injuries and deaths due to violence.

Aim 2:

1. Determine the effectiveness of complementary intervention and prevention strategies to increase interpersonal violence, substance use/disorder (IPV, SU/D), depression or anxiety screening.
2. Reduce symptoms among those who screen positive, and ultimately reduce maternal injuries and deaths due to violence.
3. Prospectively evaluate the effectiveness of a novel VIP training as the intervention condition relative to an attention control (SU/D and IPV awareness), to increase knowledge of the effects of intimate partner violence (IPV) on health outcomes, report intimate partner violence (IPV) screening behaviors, intimate partner violence (IPV) detection, and to reduce intimate partner violence (IPV) frequency among patients and clients over time.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in a helping professions program
* 18 years of age through 30 years of age
* Students whom will have direct interaction with patients or clients that may experience interpersonal violence (IPV)

Exclusion Criteria:

* Students not enrolled in a helping professions program
* Students under age 18 or over age 30
* Students with no direct interaction with patients or clients

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2800 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Knowledge and attitudes toward intimate partner violence (IPV) among pregnant and postpartum people. | Year 2 - Year 4
  Change in knowledge of intimate partner violence (IPV) and attitudes toward those experiencing IPV by condition over time. Knowledge of pregnancy-associated causes of maternal mortality and morbidity created for this randomized controlled trial (RCT). This is a 17-item scale ranging from 0-35 with higher scores indicating greater (accurate) knowledge.
Knowledge and attitudes toward substance use among pregnant and postpartum people. | Year 2 - Year 4
  Change in knowledge of substance use and attitudes toward those using substances or having a substance use disorder by condition over time. Attitudes toward pregnant or postpartum people experiencing:
  a) intimate partner violence (IPV), substance use, and anxiety or depression. This measure is based on the Domestic Violence Myth Acceptance and expanded to substance use and anxiety or depression. 45 items and 3 subscales. Response options: 1-5 indicating ranging from strongly agree to strongly disagree. Lower scores are desired indicating greater acceptance and increased willingness to address intimate partner violence (IPV), substance use, and anxiety or depression among pregnant or postpartum people.
Knowledge and attitudes toward anxiety or depression among pregnant or postpartum people. | Year 2 - Year 4
  Change in knowledge of anxiety or depression and attitudes toward those with anxiety or depression by condition over time. The Violence Against Women Health Care Provider Survey expanded to providers' willingness to ask clients about:
  a) Intimate partner violence (IPV), b) substance use, and c) anxiety or depression. 41 items querying self-confidence and actions in asking clients about risk factors for maternal morbidity. The response options 1-5 indicate strongly agree to strongly disagree. Higher scores are desired as indicators of greater self confidence and likelihood of actions with clients.

SECONDARY OUTCOMES:
Participants' (care provider) self-report of asking pregnant or postpartum people about intimate partner violence (IPV), substance use, and anxiety or depression. | Year 3 - Year 5
  Change in willingness, perceived efficacy, reports of asking clients about intimate partner violence (IPV) by condition and over time. New Bystander Action Survey developed for this randomized controlled trial (RCT). There are 20 items that measure the opportunity to take action with clients, friends or family members; actions taken, and perceived impact. There are 6 response options ranging from 0 times to more than 12 times (in the past 6 months). More actions and a higher score, are desired as indicators of greater actions to identify risk of maternal morbidity and provide resources to reduce this risk.

CONTACTS AND LOCATIONS:
Overall Officials: Ann L Coker, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official University of Kentucky website pertinent to this study — https://medicine.uky.edu/departments/obgyn/vip-corps